CLINICAL TRIAL: NCT02012543
Title: Effect of Agar Administration on Defecation and Fecal Condition in Chronic Constipated Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Showa Inan General Hospital (Other)
Responsible Party: Principal Investigator, Akira Horiuchi, Chief, Digestive Disease Center, Showa Inan General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Agar jelly; Kanten1 (Other: Ina Food Industry)
Record Dates: First submitted 2013-11-09; First posted 2013-12-16 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Constipation
Keywords: constipation, agar
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Agar jelly, constipation (Experimental): Subjects eat a cap of agar jelly (180g) shortly before eating dinner every day for 4 weeks.
  Interventions: Dietary Supplement: Agar jelly

INTERVENTIONS:
Dietary Supplement: Agar jelly

SUMMARY:
The administration of agar jelly may increase the number of defecation and the volume of feces, and then may improve fecal condition in chronic constipated patients.

DETAILED DESCRIPTION:
Each subject eats one cap of agar jelly shortly before having dinner every day for 4 weeks.

At 0, 7th, 14th, 21th, and 28th day , the frequency of defecation and defecation condition is assessed.

ELIGIBILITY:
Inclusion Criteria:

* subjects take laxatives.

Exclusion Criteria:

* subjects underwent abdominal surgery.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
the condition of feces | 4 weeks
  Bristol scale is used.

SECONDARY OUTCOMES:
the number and amount of defecation | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Akira Horiuchi, MD, Principal Investigator — Showa Inan General Hospital
Locations (1):
- Showa Inan General Hospital, Komagane, Nagano, Japan